CLINICAL TRIAL: NCT02611960
Title: A Two-arm, Open-label, Randomized Phase III Study of Pembrolizumab (MK-3475) Monotherapy Versus Standard Chemotherapy in Platinum Pre-treated, Recurrent or Metastatic Nasopharyngeal Cancer (NPC) (Keynote-122)
Brief Title: Study of Pembrolizumab (MK-3475) in Platinum Pre-treated Recurrent/Metastatic Nasopharyngeal Cancer (MK-3475-122/KEYNOTE-122)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-122; MK-3475-122 (Other: Merck); KEYNOTE-122 (Other: Merck)
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Results first posted 2021-12-15 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Capecitabine; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) until progressive disease (PD) or unacceptable toxicity for a maximum of up to 35 cycles (up to approximately 2 years). Eligible participants who stop pembrolizumab with Stable Disease (SD) or better but progress after discontinuation may be able to initiate a second course of pembrolizumab 200 mg Q3W for up to 17 cycles (up to approximately 1 additional year).
  Interventions: Biological: Pembrolizumab
- Standard Treatment (Active Comparator): Participants receive capecitabine 1000 mg/m^2 orally (PO) twice each day (BID) on Days 1-14 of each 3-week cycle, or gemcitabine 1250 mg/m^2 IV on Days 1 and 8 of each 3-week cycle, or docetaxel 75 mg/m^2 IV on Day 1 of each 3-week cycle until PD or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Gemcitabine; Drug: Docetaxel

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab
Drug: Capecitabine — oral tablet
  Other Names: XELODA®
  Arms: Standard Treatment
Drug: Gemcitabine — IV infusion
  Other Names: GEMZAR®
  Arms: Standard Treatment
Drug: Docetaxel — IV infusion
  Other Names: TAXOTERE®
  Arms: Standard Treatment

SUMMARY:
This is a study of pembrolizumab (MK-3475) versus standard treatment (capecitabine, gemcitabine, or docetaxel) for the treatment of recurrent or metastatic nasopharyngeal cancer (NPC). Participants will be randomly assigned to receive either pembrolizumab or Investigator's choice of standard treatment.

The primary study hypothesis is that pembrolizumab treatment prolongs Overall Survival (OS) when compared to standard treatment.

With Amendment 7 (effective 2-March-2022), upon study completion, participants will be discontinued and may be enrolled in an extension study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-keratinizing differentiated NPC or undifferentiated NPC
* Metastatic disease or incurable locally recurrent disease
* Treatment with prior platinum therapy
* Tumor tissue available for programmed cell death ligand 1 (PD-L1) testing
* Measurable disease based on RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* Male or female participants of childbearing potential must be willing to use an adequate method of contraception starting with the first dose of study drug through 180 days after the last dose of study drug
* Life expectancy of at least 3 months

Exclusion Criteria:

* Disease is suitable for local therapy administered with curative intent
* Participants previously treated in the recurrent/metastatic setting with any 1 of the 3 standard therapies in this study (i.e., docetaxel, capecitabine, or gemcitabine) may not receive the same therapy if randomized to the Standard Treatment arm. Additionally, participants previously treated in the recurrent/metastatic setting with all 3 standard therapies are excluded from this study
* Currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks prior to the first dose of study drug
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Not recovered from adverse events due to therapy more than 4 weeks earlier
* Prior anti-cancer monoclonal antibody (mAb) therapy within 4 weeks prior to Study Day 1, or not recovered from adverse events
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Study Day 1
* Diagnosed and/or treated additional malignancy within 5 years of randomization, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin, and/or curatively-resected in situ cervical and/or breast carcinoma
* Active autoimmune disease that has required systemic therapy in the past 2 years with modifying agents, corticosteroids, or immunosuppressive agents
* Active central nervous system metastases and/or carcinomatous meningitis
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Active infection requiring systemic therapy
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 180 days after the last dose of trial treatment for the chemotherapy arm or 120 days after the last dose of trial treatment for the pembrolizumab arm
* Prior therapy with an anti-PD-1 or anti-PD1-L1 or -L2 therapy or previously participated in a Merck pembrolizumab (MK-3475) study
* Human immunodeficiency virus (HIV) positive
* Hepatitis B or C positive
* Live vaccine within 30 days of planned start of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Chan ATC, Lee VHF, Hong RL, Ahn MJ, Chong WQ, Kim SB, Ho GF, Caguioa PB, Ngamphaiboon N, Ho C, Aziz MASA, Ng QS, Yen CJ, Soparattanapaisarn N, Ngan RK, Kho SK, Tiambeng MLA, Yun T, Sriuranpong V, Algazi AP, Cheng A, Massarelli E, Swaby RF, Saraf S, Yuan J, Siu LL. Pembrolizumab monotherapy versus chemotherapy in platinum-pretreated, recurrent or metastatic nasopharyngeal cancer (KEYNOTE-122): an open-label, randomized, phase III trial. Ann Oncol. 2023 Mar;34(3):251-261. doi: 10.1016/j.annonc.2022.12.007. Epub 2022 Dec 16. PMID 36535566
- [Derived] Chan ATC, Lee VHF, Hong RL, Ahn MJ, Chong WQ, Spreafico A, Kim SB, Ho GF, Caguioa PB, Ngamphaiboon N, Swaby RF, Wei B, Webber AL, Kang J, Gumuscu B, Yuan J, Siu LL. Analysis of Plasma Epstein-Barr Virus DNA and Clinical Outcomes to Pembrolizumab or Chemotherapy in Recurrent/Metastatic Nasopharyngeal Cancer in KEYNOTE-122. Cancer Med. 2026 Feb;15(2):e71496. doi: 10.1002/cam4.71496. PMID 41631899
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five participants randomized to the Pembrolizumab arm received a second course of pembrolizumab at the investigator's discretion as specified by the protocol. Per protocol, response/progression or adverse events (AEs) that occurred during a non-randomized second course of pembrolizumab were not counted towards efficacy or safety outcome measures, respectively. These results are for randomized treatment only.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) until progressive disease (PD) or unacceptable toxicity for a maximum of up to 35 cycles (up to approximately 2 years). Eligible participants who stopped pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab 200 mg Q3W for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Standard Treatment: Participants received capecitabine 1000 mg/m^2 orally (PO) twice each day (BID) on Days 1-14 of each 3-week cycle, or gemcitabine 1250 mg/m^2 IV on Days 1 and 8 of each 3-week cycle, or docetaxel 75 mg/m^2 IV on Day 1 of each 3-week cycle until PD or unacceptable toxicity.
Period: Overall Study
Arm/Group | Pembrolizumab | Standard Treatment
Started | 117 | 116
Discontinued | 117 | 116
Completed | 0 | 0
Not Completed | 117 | 116
Not completed — Adverse Event | 7 | 8
Not completed — Death | 98 | 92
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Sponsor Decision | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Standard Treatment | Total
Number analyzed (Participants) | 117 | 116 | 233
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.6 (12.7) | 53.1 (11.2) | 51.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 98 | 95 | 193
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 116 | 113 | 229
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 110 | 112 | 222
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 3 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Presence of Baseline Liver Metastasis [Count of Participants; unit: Participants] — The presence or absence of baseline liver metastasis(es) was reported and applied to statistical analyses. "Liver Metastasis Present" was defined as the presence of any liver metastasis and "Liver Metastasis Absent" was defined as the absence of all liver metastasis.
  Participants
    Liver Metastasis Present | 57 | 56 | 113
    Liver Metastasis Absent | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last known contact. OS was reported for each treatment arm. Per protocol, analysis for this outcome measure was performed for the first pembrolizumab course and for the standard treatment arm, with a protocol-specified analysis data cut-off date of 30-Nov-2020.
Time Frame: Up to approximately 53 months (through analysis cut-off date of 30-Nov-2020)
Population: All randomized participants (Intent-to-Treat [ITT]) were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 117 | 116
Months | 17.2 [11.7 to 22.9] | 15.3 [10.9 to 18.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Comparison based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by presence of liver metastasis; Test type: Superiority; p = 0.2262, Stratified Log-Rank Test — One-sided p-value based on log-rank test stratified by presence of liver metastasis; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.67 to 1.19]

2. Secondary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on blinded independent central review (BICR), or death due to any cause, whichever occurs earlier. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. PFS was reported for each treatment arm. Per protocol, analysis for this outcome measure was performed for the first pembrolizumab course and for the standard treatment arm, with a protocol-specified analysis data cut-off date of 30-Nov-2020.
Time Frame: Up to approximately 53 months (through analysis cut-off date of 30-Nov-2020)
Population: All randomized participants (ITT) were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 117 | 116
Months | 4.1 [2.1 to 5.6] | 5.5 [4.0 to 8.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9419, Stratified Log-Rank Test — One-sided p-value based on log-rank test stratified by presence of liver metastasis; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.94 to 1.75]

3. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1
Description: ORR was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. based upon BICR. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. ORR was reported for each treatment arm. Per protocol, analysis for this outcome measure was performed for the first pembrolizumab course and for the standard treatment arm, with a protocol-specified analysis data cut-off date of 30-Nov-2020.
Time Frame: Up to approximately 53 months (through analysis cut-off date of 30-Nov-2020)
Population: All randomized participants (ITT) were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 117 | 116
Percentage of Participants | 21.4 [14.3 to 29.9] | 23.3 [15.9 to 32.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Comparison based on Miettinen & Nurminen method stratified by presence of liver metastasis; Test type: Superiority; p = 0.63479, Stratified Miettinen and Nurminen Method — One-sided p-value for testing. H0: difference in percentage = 0 versus H1: difference in percentage > 0; Difference in Percentage = -1.9, 95% CI 2-sided [-12.7 to 8.9]

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by BICR, DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death due to any cause, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. DOR was reported for each treatment arm. Per protocol, analysis for this outcome measure was performed for the first pembrolizumab course and for the standard treatment arm, with a protocol-specified analysis data cut-off date of 30-Nov-2020.
Time Frame: Up to approximately 53 months (through analysis cut-off date of 30-Nov-2020)
Population: All randomized participants (ITT population) who demonstrated a confirmed CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 25 | 27
Months | 12.0 [6.0 to 19.9] | 13.1 [9.7 to 18.9]

5. Secondary Outcome: Percentage of Participants Surviving (OS Rate) at 12 Months
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last known contact. The percentage of participants surviving (OS rate) at 12 months is reported for each treatment arm based on the product-limit (Kaplan-Meier) method for censored data. Per protocol, analysis for this outcome measure was performed for the first pembrolizumab course and for the standard treatment arm, with a protocol-specified analysis data cut-off date of 30-Nov-2020.
Time Frame: 12 months
Population: All randomized participants (ITT) were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 117 | 116
Percentage of Participants | 58.1 [48.7 to 66.4] | 57.4 [47.8 to 65.8]

6. Secondary Outcome: Percentage of Participants Surviving (OS Rate) at 24 Months
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last known contact. The percentage of participants surviving (OS rate) at 24 months is reported for each treatment arm based on the product-limit (Kaplan-Meier) method for censored data. Per protocol, analysis for this outcome measure was performed for the first pembrolizumab course and for the standard treatment arm, with a protocol-specified analysis data cut-off date of 30-Nov-2020.
Time Frame: 24 months
Population: All randomized participants (ITT) were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 117 | 116
Percentage of Participants | 40.2 [31.3 to 48.9] | 32.2 [23.9 to 40.8]

7. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at 6 Months
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurs earlier. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. The percentage of participants with PFS (PFS rate) at 6 months is reported for each treatment arm based on the product-limit (Kaplan-Meier) method for censored data. Per protocol, analysis for this outcome measure was performed for the first pembrolizumab course and for the standard treatment arm, with a protocol-specified analysis data cut-off date of 30-Nov-2020.
Time Frame: 6 months
Population: All randomized participants (ITT) were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 117 | 116
Percentage of Participants | 36.3 [27.0 to 45.5] | 43.9 [33.6 to 53.7]

8. Secondary Outcome: Percentage of Participants With PFS (PFS Rate) at 12 Months
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurs earlier. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. The percentage of participants with PFS (PFS rate) at 12 months is reported for each treatment arm based on the product-limit (Kaplan-Meier) method for censored data. Per protocol, analysis for this outcome measure was performed for the first pembrolizumab course and for the standard treatment arm, with a protocol-specified analysis data cut-off date of 30-Nov-2020.
Time Frame: 12 months
Population: All randomized participants (ITT) were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 117 | 116
Percentage of Participants | 18.7 [11.5 to 27.3] | 30.8 [21.0 to 41.0]

9. Secondary Outcome: Percentage of Participants Who Experience One or More Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The percentage of participants that experienced at least one AE was reported for each treatment arm. Per protocol, analysis for this outcome measure was performed for the first pembrolizumab course and for the standard treatment arm.
Time Frame: Up to approximately 73 months
Population: All randomized participants who received at least 1 dose of study treatment were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 116 | 112
Percentage of Participants | 97.4 | 97.3

10. Secondary Outcome: Percentage of Participants Who Discontinue Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The percentage of participants that discontinued study treatment due to an AE was reported for each treatment arm. Per protocol, analysis for this outcome measure was performed for the first pembrolizumab course and for the standard treatment arm.
Time Frame: Up to approximately 72 months
Population: All randomized participants who received at least 1 dose of study treatment were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 116 | 112
Percentage of Participants | 8.6 | 15.2

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events (including first and second courses): Up to approximately 73 months (through Final Analysis cut-off date of 30-Sep-2022)
Description: All-Cause Mortality table includes all randomized participants. Serious and Other AEs include all treated participants according to treatment received. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" unrelated to drug were excluded as AEs. Five participants randomized to Pembrolizumab arm received a second course of pembrolizumab per protocol and were monitored for AEs and All-Cause Mortality separately.
Groups:
- Pembrolizumab First Course: Participants received pembrolizumab 200 mg IV Q3W until PD or unacceptable toxicity for a maximum of up to 35 cycles (up to approximately 2 years).
- Standard Treatment First Course: Participants received capecitabine 1000 mg/m^2 orally (PO) twice each day (BID) on Days 1-14 of each 3-week cycle, or gemcitabine 1250 mg/m^2 IV on Days 1 and 8 of each 3-week cycle, or docetaxel 75 mg/m^2 IV on Day 1 of each 3-week cycle until PD or unacceptable toxicity.
- Pembrolizumab Second Course: Eligible participants randomized to the pembrolizumab arm who stopped pembrolizumab with SD or better but progressed after discontinuation initiated a second course of pembrolizumab at the investigator's discretion at the same dose and schedule (200 mg Q3W) for up to 17 cycles (up to approximately 1 additional year).
Arm/Group | Pembrolizumab First Course | Standard Treatment First Course | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 103/117 | 104/116 | 3/5
Serious Adverse Events (participants affected / at risk) | 39/116 | 41/112 | 3/5
Other Adverse Events (participants affected / at risk) | 100/116 | 103/112 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=116) | Standard Treatment First Course (N=112) | Pembrolizumab Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 9 (10) | 9 (10) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 4 (7) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (6) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=116) | Standard Treatment First Course (N=112) | Pembrolizumab Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 13 (15) | 33 (47) | 0 (0)
Hypothyroidism (Endocrine disorders) | 20 (20) | 11 (12) | 0 (0)
Vision blurred (Eye disorders) | 6 (6) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (8) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 13 (15) | 17 (20) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (17) | 19 (27) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 6 (7) | 4 (7) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 8 (10) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (12) | 18 (30) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 16 (19) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (21) | 17 (20) | 0 (0)
Chest pain (General disorders) | 10 (12) | 2 (2) | 0 (0)
Chills (General disorders) | 5 (11) | 6 (8) | 0 (0)
Fatigue (General disorders) | 24 (29) | 29 (37) | 0 (0)
Malaise (General disorders) | 7 (9) | 6 (7) | 0 (0)
Mucosal inflammation (General disorders) | 3 (4) | 10 (13) | 0 (0)
Oedema peripheral (General disorders) | 6 (7) | 7 (8) | 0 (0)
Pyrexia (General disorders) | 18 (29) | 28 (51) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (8) | 8 (13) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 13 (17) | 16 (24) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (9) | 5 (13) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 10 (10) | 5 (8) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 9 (10) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 5 (6) | 11 (14) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 38 (109) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 10 (61) | 0 (0)
Weight decreased (Investigations) | 8 (9) | 7 (7) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 19 (52) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 23 (24) | 14 (18) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (17) | 8 (20) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (13) | 7 (11) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (22) | 4 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (16) | 13 (15) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 9 (10) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (12) | 5 (7) | 0 (0)
Dizziness (Nervous system disorders) | 16 (21) | 20 (22) | 0 (0)
Headache (Nervous system disorders) | 16 (19) | 11 (22) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 6 (6) | 4 (4) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 8 (9) | 0 (0)
Insomnia (Psychiatric disorders) | 13 (14) | 11 (13) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 34 (51) | 19 (32) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 5 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 13 (20) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 11 (14) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (11) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 11 (15) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 16 (17) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 9 (9) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 22 (28) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (22) | 13 (16) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 20 (32) | 20 (30) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 12 (13) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT02611960/Prot_SAP_001.pdf